CLINICAL TRIAL: NCT04780048
Title: Complex Abdominal Wall Reconstruction Using Biologic Mesh Outcomes Prospective Study
Brief Title: Complex Abdominal Wall Reconstruction Using Biologic Mesh
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Rifat Latifi, Professor, General surgery, New York Medical College
Other Study IDs: L#12086
Record Dates: First submitted 2020-08-13; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Hernia
Keywords: Hernia repair
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine how the patient factors, co-morbid conditions, pre-operative workup, anatomy of the defect, reconstruction details, operative techniques, and type of repairs contribute to the final outcome of abdominal wall reconstruction. The outcomes of interest are: in-hospital complications, discharge disposition, hospital and ICU length of stay, long term follow-up (recurrence, reoperation, and explantation rates).

DETAILED DESCRIPTION:
Background:

Abdominal wall defects are commonly seen in trauma and EGS patients. During the last decade numerous advances have been made in the management of patients with abdominal wall defects. These defects are repaired by various surgical techniques including mesh repair (synthetic vs. biologic), primary repair, etc. However, the outcomes of patients after these injuries are highly variable and many of these patients suffer from in-hospital complications, mesh infections requiring explantation, and recurrence. Various factors play a role in the final outcome of the patient. These include factors associated with the initial surgery or disease (trauma or emergency general surgery), patient demographics (age, gender, co-morbidities), preoperative features (hemoglobin and laboratory parameters), technique of repair (onlay, inlay, retro rectus) and the types of mesh used. However, the role of each of these factors in the final outcome of patients remains unclear in the literature.

Study Design Study Type: Observational Observational Study Model: Cohort Time Perspective: Prospective Enrollment: 250 Number of Groups/Cohorts: 1

Recruitment Procedures:

Attending physicians will discuss possible participation in the study with patients who meet initial screening criteria and have been scheduled for abdominal wall repair/ventral hernia repair. If a patient agrees, they will be approached by our research coordinator to discuss consenting. The research coordinator will introduce herself and her role with Westchester Medical Center, and read the following script. A translator for Spanish speaking patients will be available.

Hello, my name is _______________. I am a research coordinator with the Department of Surgery here at Westchester Medical Center. I'm talking to you today because you or your family member are scheduled to have a surgery that involves abdominal wall repair. Dr. Latifi, the Director of the Department of Surgery, is conducting a study looking at outcomes from this surgery. We are interested in how this procedure and personal factors, such as having diabetes, may contribute to how long you stay in the hospital, have a recurrence or develop an infection. Participation in this study does not require anything additional from you. You will receive the same care if you do or do not participate. The only difference is we would maintain your outcome data for analysis purposes. Would you be interested in learning more about the study and discussing study details with me and Dr. Latifi? If so, are you able to meet and when would you like to meet? Or, if you do not know yet, can you provide me with your phone number or the best way to contact you to schedule a follow-up meeting to discuss the study?

Research Coordinator meets and collects potential participant contact information.

Meeting will be held to describe study in more detail and to consent participant and/or representative. If participant is already in the hospital for the procedure, the meeting will be held as soon as possible.

Data management:

The research involves no more than minimal risk to subjects as it provides no additional treatment for patients who had abdominal wall defects and are undergoing surgery. Data will be obtained on their pre and perioperative details, their interventions, and final outcomes. This study will use a chart review of data from electronic medical records for current patients. Subjects will be recruited, consented, and medical record data will be gathered prospectively.

Medical records containing Protective Health Information such as admission and discharge date will be obtained from the hospital Electronic Medical Record database in the form of a query spreadsheet to determine hospital and ICU length of stay. All data will be de-identified using a unique identifier that is assigned to each record.

Data will be queried from the database and kept in a password protected excel spreadsheet. Only the PI and designated research personnel will have the access to the Protective Health Information and data linkage file. The PI designated research team members will have the access to the de-identified data.

Data will be stored and secured in a logbook/secured computer with the PI. Hard copies will also be stored in closed envelopes in locked cabinets in PI's office. The data will be kept for a period of seven years and then later will be destroyed. Data will be stored by the Westchester Medical Center (WMC) Lead PI.

Analytic Plan: Chi-square difference tests will be used to assess significant differences in predictors on categorical outcomes. T-tests will be used to assess mean differences in predictors on continuous outcomes. Univariable and multivariable logistic regression analyses will be conducted for outcomes such as all-cause mortality, pneumonia, sepsis, and multi-organ failure. Univariable and multivariable linear regression will be performed for hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

• All patients aged 18 years and above undergoing Abdominal wall reconstruction with biological mesh.

Exclusion Criteria:

• Vulnerable patient population (Neonates, Prisoners, Pregnant) will not be included in our study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 years and above undergoing Abdominal wall reconstruction with biological mesh irrespective of gender, ethnicity, socio-economic status will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2022-07-06 (Estimated); Study Completion 2022-12-06 (Estimated)

PRIMARY OUTCOMES:
In Hospital Complications | 3 years
  Infection, re-procedures, explantation rates, length of hospital stay and ICU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Rifat Latifi, MD, Principal Investigator — Chairman Department of Surgery
Locations (1):
- Westchester Medical center, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
no plans